CLINICAL TRIAL: NCT04050137
Title: Therapeutic Exercise to Treat Neuropathic Pain in Patients With Chronic Lisosomal Injuries: Learning and Service Project
Brief Title: Therapeutic Exercise to Treat Neuropathic Pain
Acronym: Aps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: fundación española para el estudio y tratamiento de la Enfermedad de Gaucher y otras lisosomales (Unknown); Fundación San Valero (Unknown); Fundación Ibercaja (Unknown)
Responsible Party: Principal Investigator, Maria Pilar López Royo, Principal Investigator, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI19/205
Record Dates: First submitted 2019-04-23; First posted 2019-08-08 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Gaucher Disease; Fabry Disease
Keywords: Gaucher Disease; Exercise; Terapheutic
MeSH Terms: conditions — Gaucher Disease; Fabry Disease; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Exercise programme 3 times/week.
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Other: Therapeutic Exercise — Patients who meet the inclusion criteria and who want to carry out the workshops, fill out an informed consent explaining the procedure to be followed and accepting the cessation of data to carry out the study.
  Patients will be divided into 2 working groups (approximately 10 patients in total, in a Gaucher disease group and in another Fabry disease). The workshops will be held at the foundation twice a month in sessions of 45 minutes of work for 3 months (May, June, July 2019). In these sessions the physiotherapists will show the new exercises to the patients. The exercises that are taught in that session should be done at home 3 times a week. In addition, a document will be delivered with the exercises to be carried out and the frequency and intensity of execution. The workshops will be guided at all times by a physiotherapist specialized in therapeutic exercise and EDL.

SUMMARY:
A quasi-experimental, prospective clinical trial with pre and post intervention measurements, whose porpuose is assess the efficacy of a therapeutic exercise protocol to treat neuropathic pain in Fabry Disease.

DETAILED DESCRIPTION:
There take part in this study women or men aged between 18 and 65 years, with a diagnosys by a physician specializing in Fabry disease with FabryScan. Patients must present a stable evolution, with a scoring system of disease severity (DS3) that must be less than 8 points per year in the last 2-3 years and they have to presence of neuropathic pain with a score greater than or equal to 4 in the questionnaire "Douleur neuropathique (DN4)".

ELIGIBILITY:
Inclusion criteria:

* Female or male patients between 18 years and 65 years.
* Patients diagnosed by a doctor specializing in Fabry disease with FabryScan.
* Fabry's disease must have a stable evolution, with a disease severity scoring system (DS3) that must be less than 8 points per year in the last 2-3 years.
* Presence of neuropathic pain with a score greater than or equal to 4 in the "Douleur neuropathique (DN4)" questionnaire.

Exclusion criteria:

* Patients with an acute cardiovascular disease or with a heart or kidney transplant.
* Subjects with acute orthopedic problems that limit their participation in the study.
* Subjects with cognitive impairments that prevent them from filling in the questionnaires or understanding the exercises to be performed.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Neurophatic pain | 8 weeks
  DN4. This tool allows to estimate the probability of neuropathic pain of the patient in a valid and reliable way. It consists of 4 questions with 10 items to fill out. The researcher directly asks the patient and it is the investigator who completes the questionnaire. To each item, you must provide a "yes" or "no" answer; the "yes" is worth 1 point and the "no" is worth 0 point. At the end of the questionnaire, the investigator counts the patient's score on 10. If the patient's score is equal to or greater than 4 out of 10, the test is positive.

SECONDARY OUTCOMES:
Functionality | 8 weeks
  Arm Functionality DASH. The DASH questionnaire is a tool for assessing and measuring the functionality of the upper limb that the patient perceives during daily activities. This questionnaire is used in several studies with patients with disabilities in the hand, elbow and shoulder. It is valid, reliable and capable of detecting changes.
Legs' strenght | 8 weeks
  Test of rising and sitting of the chair during 30 seconds as many times as possible.
Strenght of the extensor muscless of the trunk | 8 weeks
  BST. Biering-Sorensen test.The test is to keep the trunk in prone position as long as possible to assess the resistance of the trunk extensor musculature.
Strenght of the inclination muscless of the trunk | 8 weeks
  TSB. Test Side-Bridge assesses the resistance of the inclination muscles or lateral flexors of the trunk. In it the participants are placed in lateral recumbency on their dominant side in a mat. In this position, the participants support themselves with the elbow and the forearm of their dominant side and raise the pelvis until the trunk is aligned with the lower extremities. The test consists of maintaining the referred position as long as possible.
Strenght of the flexor muscless of the trunk | 8 weeks
  ITo. To assess the resistance of the flexor muscles of the trunk, the participants are placed supine with the hips and knees bent at 90º. The participants flex the upper part of the trunk until they touch the thighs with the elbows, keeping the cervical spine in a neutral position.
Visual Analogue Scale | 8 weeks
  VAS. The analog visual pain scale is a tool that is used to assess the pain perceived by the patient in a valid and reliable way.
  It is an instrument for measuring the intensity of pain that represents a horizontal line of 10 cm with a score of 0 to 10, where 0 represents non-pain and 10 unbearable pain.
  The patient should place a vertical line on the horizontal line of the scale where he places his pain intensity.
Hospital, anxiety and depression questionnaire | 8 weeks
  HADS. This questionnaire allows to evaluate the psychosocial factors of the patient, through 14 questions with two subscales of 7 questions (one subscale on anxiety and the other on depression); The patient must answer one of the 4 items of each question without much reflection to have a real answer of how he was during the past week. The intensity or frequency of symptoms is evaluated with a Likert scale ranging from 0 to 3. In each subscale (anxiety and depression) the points are added and interpreted as such: 0-7 points: normal; 8-10 points: doubtful and higher than 11: clinical problem. This tool is validly and reliably used in clinical practice.
SF-36 | 8 weeks
  This questionnaire assesses the quality of life perceived by the patient. It is widely used in clinical practice and is approved as valid and reliable. There are 36 questions with 2,3,5 or 6 items in each question and with an assessment between 0 and 100. The questions assess physical function, function limitations due to physical health problems, body aches, general health, vitality, social functioning and emotional and mental health problems
Semmes Weinstein monofilament test | 8 weeks
  The Semmes Weinstein monofilament test is a tool that evaluates tactile and pressure sensitivity in a valid and reliable way. A nylon filament attached to a handle is used which, when folded, applies a constant pressure of 10g. The investigator applies the monofilament perpendicular to the skin with increased pressure until the monofilament bends and without supporting it for more than 1 or 2 seconds.
  The test will be performed on the sole of the foot in 4 points: the first toe, the base of the first, third and fifth metatarsals.
  When the patient notices something, he puts a 1 and a 0 if he does not notice something. The sensitivity index is obtained with the sum of the values and is considered a sensitive patient only when it has a score of 8/8.

CONTACTS AND LOCATIONS:
Overall Officials: Royo, Principal Investigator — Universidad San Jorge
Locations (1):
- FEETEG, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No